CLINICAL TRIAL: NCT02609451
Title: Closure of Protective Ileostomy 2 vs. 12 Weeks Following Total Mesorectal Excision (TME) for Rectal Surgery: Interim Analysis of a Multicentre, Randomized, Controlled Study
Brief Title: Closure of Protective Ileostomy 2 vs. 12 Weeks After TME
Acronym: Closure2vs12
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Evidence of bad outcome after interims analysis
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKBB-REF-NR-266/07_Ileostomy
Record Dates: First submitted 2015-09-24; First posted 2015-11-20 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-01

CONDITIONS: Rectal Cancer
Keywords: quality of life; feasibility; safety; protective ileostomy closure
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 weeks (Experimental): Ileostomy closure after 2 weeks
  Interventions: Procedure: Ileostomy closure
- 12 weeks (Experimental): Ileostomy closure after 12 weeks
  Interventions: Procedure: Ileostomy closure

INTERVENTIONS:
Procedure: Ileostomy closure — Ileostomy closure at a different time point

SUMMARY:
The purpose of this study is to compare the feasibility, safety, and quality of life (QOL) in patients (pts) undergoing protective ileostomy closure after 2 weeks with a closure after 12 weeks.

DETAILED DESCRIPTION:
In three surgical departments between 2007 and 2013, 72 pts with total mesorectal excision and coloanal or low colorectal anastomosis for rectal cancer were randomly assigned to closure of their protective ileostomy after 2 weeks (group A, 37 pts) or 12 weeks (group B, 35 pts). One day before planned stoma closure, the coloanal/colorectal anastomosis was checked by palpation, contrast enema via ileostomy and, in case of hazards, by proctoscopy. Perioperative data was assessed prospectively using numeric values, visual analogue scales (VAS, 0 = lowest value, 100 = highest value) and QOL-index (GQLI, max. 144 points). Complications were recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

* anastomosis ≤ 5cm from anal verge
* age >18 years
* informed consent
* uneventful course after first operation

Exclusion Criteria:

* pregnancy
* allergy to contrast agent
* severe non-surgical complications
* evident abdominal - pelvic complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Quality Of Life (GQLI - Questionnaire) | 6 weeks
  Quality Of Life Survey using the GQLI - Questionnaire

SECONDARY OUTCOMES:
Feasibility (via Visual Analogue Scale) | intraoperatively
  Surgical Feasibility including blood loss, blood oozing, epifascial and intrabdominal adhesions, operating time and difference in bowel diameter
Safety as assessed by Morbidity, Mortality | 6 weeks, 16 weeks
  Morbidity, Mortality
Quality Of Life (EORTC - Questionnaire) | preoperative (preOP), 6 weeks, 16 weeks
  Quality Of Life Survey using the EORTC - QLQ C30 - Questionnaire
Quality Of Life (GQLI - Questionnaire) | preOP, 16 weeks
  Quality Of Life Survey using the GQLI - Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A. Maurer, Prof.Dr.med., Principal Investigator — Cantonal Hosptal, Baselland
Locations (1):
- Kantonspital Baselland Liestal, Liestal, Basel-Landschaft, Switzerland

REFERENCES:
- [Background] Thalheimer A, Bueter M, Kortuem M, Thiede A, Meyer D. Morbidity of temporary loop ileostomy in patients with colorectal cancer. Dis Colon Rectum. 2006 Jul;49(7):1011-7. doi: 10.1007/s10350-006-0541-2. PMID 16598401
- [Background] O'Leary DP, Fide CJ, Foy C, Lucarotti ME. Quality of life after low anterior resection with total mesorectal excision and temporary loop ileostomy for rectal carcinoma. Br J Surg. 2001 Sep;88(9):1216-20. doi: 10.1046/j.0007-1323.2001.01862.x. PMID 11531870
- [Background] Hallbook O, Matthiessen P, Leinskold T, Nystrom PO, Sjodahl R. Safety of the temporary loop ileostomy. Colorectal Dis. 2002 Sep;4(5):361-364. doi: 10.1046/j.1463-1318.2002.00398.x. PMID 12780582
- [Derived] Elsner AT, Brosi P, Walensi M, Uhlmann M, Egger B, Glaser C, Maurer CA. Closure of Temporary Ileostomy 2 Versus 12 Weeks After Rectal Resection for Cancer: A Word of Caution From a Prospective, Randomized Controlled Multicenter Trial. Dis Colon Rectum. 2021 Nov 1;64(11):1398-1406. doi: 10.1097/DCR.0000000000002182. PMID 34343161